CLINICAL TRIAL: NCT06441513
Title: The Preventive Effect of Chinese Traditional Medicine Nursing Combined With Case Tracking Management on Chemotherapy-induced Hand-foot Syndrome: a Randomized Controlled Study
Brief Title: The Preventive Effect of Chemotherapy-induced Hand-foot Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Chen Yamei, Head nurse, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LM2023104
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: Hand foot syndrome; Case Tracking management; TCM External Treatment Nursing
MeSH Terms: conditions — Neoplasms; Hand-Foot Syndrome

STUDY DESIGN:
Intervention Model Description: The process of randomization and concealment allocation was conducted by a research team who were not involved in the study. Spss26.0 software was used to program and generate a random number table, which was randomly divided into two groups.
Who Masked: Outcomes Assessor
Masking Description: Random numbers were sequentially sealed in a continuously numbered and opaque envelope. The envelopes were opened sequentially to allocate participants to the case tracking management or control group by the other researcher. Because of the nature of continuing care intervention, it was not possible to blind the participants about the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invention group (Experimental): On the basis of the intervention measures in the control group, we added the following measures. First, we set up a team for the prevention of hand foot syndrome, including 1 head nurse of the tumor chemotherapy department, 2 doctors, 16 nurses (16 nurses were divided into 4 groups, each group designated a team leader) and the researchers of this experiment. Doctors are responsible for the diagnosis of HFS and the determination of traditional Chinese medicine prescriptions, head nurses and team leaders are responsible for quality control, and nurses are responsible for the assessment, intervention and evaluation of patients.
  Interventions: Other: Chinese traditional medicine nursing combined with case tracking management
- Control group (Other): We distributed traditional Chinese medicine to the control group and carried out health education, which mainly included elaborating the symptoms, mechanism and corresponding treatment measures of HFS for patients, reducing the fear of patients, helping them relax and adjust their mentality, and cooperating with observation. At the same time, we should also try to reduce the chance of skin damage on hands / feet, such as wearing long clothes and pants when going out to avoid direct sunlight; Wear loose shoes, socks and gloves to avoid frequent friction and excessive pressure of hands and feet; Avoid heavy physical labor and intense exercise; Avoid contact with supercooled, overheated, sharp and irritating objects.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Chinese traditional medicine nursing combined with case tracking management — First, we set up a team for the prevention of hand foot syndrome, including 1 head nurse of the tumor chemotherapy department, 2 doctors, 16 nurses (16 nurses were divided into 4 groups, each group designated a team leader) and the researchers of this experiment. Doctors are responsible for the diagnosis of HFS and the determination of traditional Chinese medicine prescriptions, head nurses and team leaders are responsible for quality control, and nurses are responsible for the assessment, intervention and evaluation of patients.
  Other Names: Health Education
  Arms: Invention group
Other: Health Education — elaborating the symptoms, mechanism and corresponding treatment measures of HFS for patients, reducing the fear of patients, helping them relax and adjust their mentality, and cooperating with observation.
  Arms: Control group

SUMMARY:
this study will use traditional Chinese medicine bath with no obvious side effects combined with case tracking management mode to form nursing measures to prevent hand foot syndrome. A randomized controlled trial design will be used to collect cases of hand foot syndrome (HFS) that did not appear after chemotherapy in the ward of the Department of chemotherapy, Peking University Third Hospital, and carry out nursing intervention.

DETAILED DESCRIPTION:
Chemotherapy drugs have achieved certain satisfactory clinical efficacy in the treatment of cancer, but they can also cause common side effects including digestive tract reactions, skin rashes, hand-foot syndrome, and bone marrow suppression. Among them, hand-foot syndrome (HFS) is a common chemotherapy complication with an incidence rate of up to 50%-60%6. About 17%-24% of patients may develop grade 3 HFS. The main clinical manifestation of HFS is characterized by red plaques and sensory abnormalities on the palms and soles of the hands and feet. The initial symptoms are hyperemia and erythema on the palms and soles, tingling sensation, sensory abnormalities/sensory insensitivity, numbness at the ends of the fingers/toes, followed by tension, pain, dryness, skin desquamation and peeling (small or large flakes of skin lifted) on the hands and feet. In severe cases, blisters, exudation, and even ulcers may occur, accompanied by severe pain. Patients may be unable to walk or hold objects due to pain, and even lose their ability to take care of themselves. Currently, HFS is mainly treated by interrupting chemotherapy, symptomatic analgesia, anti-inflammation, and preventing infection. The occurrence of HFS brings great inconvenience to patients' daily lives, not only affecting their ability to live independently (including general labor and work), but also adding additional economic expenses. More importantly, due to the impact of drug reduction or withdrawal, cancer treatment cannot be carried out smoothly, which has a negative impact on patients' quality of life. Therefore, paying attention to the prevention of hand-foot syndrome is of great clinical significance.

At present, domestic and foreign scholars have adopted oral administration of vitamin, mecobalamin and other neuroprotective drugs to prevent HFS， but the incidence of HFS remains high. The analysis of the reasons found that due to the lack of effective management, patients have poor compliance, and patients are worried about the side effects of drugs, which further reduces their compliance. Many domestic studies have found that external treatment of traditional Chinese medicine (including bathing and application) is safe, effective and easy to implement. Moreover, more and more studies have found that traditional Chinese medicine can effectively treat hand-foot syndrome Case tracking management mode is a branch of tracking methodology, which refers to tracking the diagnosis, treatment and nursing process experienced by patients in the whole medical system, evaluating the nursing service of the hospital from the perspective of "patients", so that the evaluator can "see" the whole nursing process from the perspective of patients. In recent years, studies have found that the case tracking management model can quickly find and improve the quality of clinical nursing problems, and has a significant role in promoting high-quality nursing and nursing safety. Therefore, this study will use traditional Chinese medicine bath with no obvious side effects combined with case tracking management mode to form nursing measures to prevent hand foot syndrome. A randomized controlled trial design will be used to collect cases of hand foot syndrome (HFS) that did not appear after chemotherapy in the ward of the Department of chemotherapy, Peking University Third Hospital, and carry out nursing intervention.

ELIGIBILITY:
Inclusion Criteria:

* (1) no HFS symptoms in chemotherapy patients; (2) Ages 18 to 65 years; (3) Estimated survival ≥ 3 months; (4) There was no dysfunction of major organs, heart, liver and kidney functions were basically normal, and the laboratory indicators met the following requirements: neutrophils > 1.5 × 109/l, platelets > 100 × 109/l, hemoglobin > 90g/l; Bilirubin was normal or < 1.5 × ULN; AST and alt < 2.5 × ULN; Serum creatinine < 1.5 × ULN; Endogenous creatinine clearance (CCR) ≥ 60ml/min. (5) Those who can understand the situation of this study, can cooperate in the assessment of HFS grading, and have signed the informed consent.

Exclusion Criteria:

* (1) history of nerve trauma before chemotherapy, diabetic neuropathy, spinal cord compression syndrome without surgical treatment, spinal canal stenosis or spinal cord nerve root compression, and central nervous system tumors; (2) Patients with skin lesions of hands and feet; (3) Those who have plans to use other drugs that may affect HFS (including urea cream, vitamin B6, celecoxib, compound Sophora flavescens injection, calf blood deproteinized extract intravenous injection); (4) Patients with severe, uncontrolled organic lesions or infections, such as decompensated heart, lung, renal failure, etc., that lead to intolerance to chemotherapy; (5) Those who participate in other clinical trials at present or within 4 weeks; (6) Obvious neurological and psychiatric history, including dementia or epilepsy that may affect understanding and informed consent; (7) Intolerant or allergic to the traditional Chinese medicine prescriptions in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of HFS | At the end of 42 days of chemotherapy for the patient
  Number of HFS patients / total number of patients included in each group

SECONDARY OUTCOMES:
EORTC-QOL-C30 | At the end of 42 days of chemotherapy for the patient
  QoL was measured by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire （EORTC-QOL-C30）

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Chen, Study Chair — Peking University Third Hospital Library
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on reasonable request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Miller KK, Gorcey L, McLellan BN. Chemotherapy-induced hand-foot syndrome and nail changes: a review of clinical presentation, etiology, pathogenesis, and management. J Am Acad Dermatol. 2014 Oct;71(4):787-94. doi: 10.1016/j.jaad.2014.03.019. Epub 2014 May 1. PMID 24795111
- [Result] Kanbayashi Y, Taguchi T, Ishikawa T, Otsuji E, Takayama K. Risk Factors of Capecitabine-Induced Hand-Foot Syndrome: A Single-Institution, Retrospective Study. Oncology. 2023;101(7):407-414. doi: 10.1159/000529851. Epub 2023 Apr 19. PMID 37075722
- [Result] Kao YS, Lo CH, Tu YK, Hung CH. Pharmacological prevention strategy for capecitabine-induced hand-foot syndrome: A network meta-analysis of randomized control trials. Dermatol Ther. 2022 Oct;35(10):e15774. doi: 10.1111/dth.15774. Epub 2022 Aug 30. PMID 36054263